CLINICAL TRIAL: NCT00378196
Title: Ranibizumab in Idiopathic Parafoveal Telangiectasia (RIPT) Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Neil M. Bressler, Principal Investigator, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00002686
Record Dates: First submitted 2006-09-18; First posted 2006-09-19 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Telangiectasia
Keywords: Idiopathic Parafoveal Telangiectasia (IPT); Also Known As Idiopathic Juxtafoveal Telangiectasia (IJFT)
MeSH Terms: conditions — Telangiectasis | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): 0.3 mg/0.05 ml dose of ranibizumab
  Interventions: Drug: Ranibizumab
- B (Experimental): 0.5 mg /0.05 ml dose of ranibizumab
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — 0.3 mg/0.05 ml dose
  Other Names: Lucentis
  Arms: A
Drug: Ranibizumab — 0.5 mg/0.05 ml dose
  Other Names: Lucentis
  Arms: B

SUMMARY:
This research is being done to look at the effects of an experimental drug, ranibizumab, for the treatment of a condition called "idiopathic parafoveal telangiectasia" or IPT. IPT is caused by swelling in the retina (the light sensitive tissue in the back of the eye) due to leaky blood vessels in this area. Swelling in the retina can lead to blurry vision.

DETAILED DESCRIPTION:
This study is a randomized, interventional case series. A total of 10 patients, seen in the Retina Division of the Wilmer Eye Institute, will be enrolled. Subjects will be randomized to either 0.3 mg or 0.5 mg intravitreal injections of ranibizumab. Patients with IPT with macular edema documented on optical coherence tomography (OCT) but no choroidal neovascularization will be eligible for this study. Exclusion criteria will include other forms of retinopathy, active intraocular inflammation, history of poor vision due to conditions other than IPT in either eye, and known hypersensitivity to humanized monoclonal antibodies.

After obtaining informed consent, the patient will undergo baseline assessment including best-corrected Early Treatment for Diabetic Retinopathy Study (ETDRS) visual acuity, ocular examination, color fundus photography, fluorescein angiography, and OCT. If both eyes are eligible, the study participant and investigator will choose which eye to be considered the study eye. The study eye will be assigned at random to receive an intravitreal dose of ranibizumab (0.3 mg/0.05 ml or 0.5 mg/0.05 ml) at the baseline, 1 month, and 2 month visits. Further monthly injections are at the discretion of the examiner, and may be withheld if there is lack of continued improvement (defined as lack of improvement of at least 5 letters on an eye chart compared with 2 previous consecutive visits or lack of decrease of the retinal center point thickness of at least 50 microns compared with 2 previous consecutive visits) or complete success (defined as visual acuity of 20/20 or better or retinal center point thickness <225 microns).

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible if the following criteria are met:

  1. Ability to provide written informed consent and comply with study assessments for the full duration of the study.
  2. Age > 18 years
  3. Diagnosis of bilateral IPT with macular edema documented on OCT and no evidence of choroidal neovascularization.
  4. Best corrected visual acuity of better or equal to 20/200 in both eye

Exclusion Criteria:

* Subjects who meet any of the following criteria will be excluded from this study:

  1. Known hypersensitivity to humanized monoclonal antibodies
  2. History (within past 6 months) or evidence of severe cardiac disease (apparent in electrocardiogram abnormalities, clinical history of unstable angina, acute coronary syndrome, myocardial infarction, revascularization procedure within 6 months prior to baseline, atrial or ventricular tachyarrhythmias requiring ongoing treatment).
  3. History of stroke within 6 months of study entry.
  4. Current acute ocular or periocular infection.
  5. Any major surgical procedure within one month of study entry.
  6. Known serious allergies to fluorescein dye.
  7. Previous participation in a clinical trial (for either eye) involving anti-angiogenic drugs (pegaptanib, ranibizumab, anecortave acetate, Protein Kinase C inhibitors, etc) within last 6 months.
  8. Previous intravitreal drug delivery (e.g., intravitreal corticosteroid injection or device implantation) in the study eye within the last 6 months.
  9. History of subfoveal laser treatment in the study eye.
  10. History of other visually-limiting conditions such as optic neuropathy, amblyopia, choroidal neovascularization due to causes other than IPT in the study eye.
  11. Ocular inflammation (including trace or above) in the study eye.
  12. Inability to comply with study or follow up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-09; Primary Completion 2007-09 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with improvement of 15 or more letters of best corrected visual acuity from baseline to 3 months on an Early Treatment Diabetic Retinopathy visual acuity chart measured at 4 meters | 3 months

SECONDARY OUTCOMES:
Retinal changes on ophthalmoscopy | 3 months
Retinal thickness measured by Optical Coherence Topography (OCT) | 3 months
Fluorescein leakage on fluorescein angiography | 3 months
Complications related to drug or its administration | 12 months after last injection

CONTACTS AND LOCATIONS:
Overall Officials: Neil M. Bressler, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Wilmer Eye Institute at Johns Hopkins, Baltimore, Maryland, United States